CLINICAL TRIAL: NCT00086398
Title: Psychotherapy Enhancement for TC Retention
Brief Title: Psychotherapy Enhancement for Therapeutic Community (TC) Retention - 1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Model: Factorial | Purpose: Treatment
Other Study IDs: NIDA-14967-1; R01-14967-1
Record Dates: First submitted 2004-07-01; First posted 2004-07-07 (Estimated); Last update posted 2005-11-07 (Estimated); Status verified 2005-11

CONDITIONS: Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Behavior Therapy

INTERVENTIONS:
Behavioral: Behavior Therapy

SUMMARY:
The purpose of this study is to evaluate the efficacy of Dual Focus Schema Therapy in comparison to Individual Drug Counseling as 6-month manualized individual behavioral therapy enhancements to the orientation/early treatment process of Therapeutic Community (TC) residents.

DETAILED DESCRIPTION:
Therapeutic Community (TC) treatment can be effective psychosocial modality for addiction, but premature dropout remains a major problem. Personality disorders are very common in residential programs, and TCs regard personality disturbance as core to all people with addiction. Severe personality dysfunction is associated with higher dropout rates from TCs, and adding cognitive-behavioral treatments may improve retention and outcome. We hypothesize that severe personality disturbance causes significant problems with an individual?s initial adjustment and effective utilization of TC processes and techniques. We predict that a behavioral therapy that targets personality pathology will result in better early retention and engagement than will a more standard addiction counseling approach.

To begin to improve retention, TC research must begin to systematically evaluate the impact of adding interventions targeted at decreasing premature dropouts through controlled clinical trials. We have developed the first empirically tested treatment manual for the full range of personality disorders in substance abusers and propose to conduct a randomized clinical trial to evaluate the efficacy of Dual Focus Schema Therapy in comparison to Individual Drug Counseling as 6-month manualized individual behavioral therapy enhancements to the orientation/early treatment process of 100 TC residents. In addition to evaluating retention differences, we will analyze the rate and degree of change for these two conditions monthly and at 6, 12, 18, and 24-month follow-up for psychological indicators related to personality disorder and therapeutic processes related to the TC.

ELIGIBILITY:
Admission for residential TC treatment at APT Residential Services Division

Inclusion Criteria:

Adolescent or adult substance abuser; provide 2 or more contacts; ability to read and speak English

Exclusion Criteria:

Acute suicidality, homicidality, psychosis, mania

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2001-09

PRIMARY OUTCOMES:
Retention
Psychosocial functioning

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Ball, Ph.D., Principal Investigator — APT Foundation, Inc.
Locations (1):
- APT Residential Services Division, New Haven, Connecticut, United States